CLINICAL TRIAL: NCT04299191
Title: Study of LAM561 Acid in Pediatric Patients With Malignant Glioma and Other Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Laminar Pharmaceuticals (Industry)
Collaborators: Hackensack Meridian Health (Other); Dana-Farber Cancer Institute (Other); Laminar Pharma Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MIN-001P-1501
Record Dates: First submitted 2020-02-25; First posted 2020-03-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: High-grade Glioma; Solid Tumor, Unspecified, Child
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Intervention Model Description: An open label, non-randomized study in pediatric patients with advanced high-grade gliomas and other solid tumors.
  The study will be performed in two phases: a dose escalation phase in up to 18 patients following a standard "3+3" design to establish dose-limiting toxicity (DLT) and a "safe" dose of LAM561 followed by an expanded safety cohort of up to 10 patients treated at the Maximum Tolerated Dose (MTD). If the MTD is well tolerated in the expanded safety cohort, that dose becomes the Recommended Phase 2 Dose (RP2D).
  Glioma patients and other solid tumor patients (including non-glial brain tumors) will be treated as a single cohort. Patients with either tumor type will be allowed to enroll on the study as positions are made available. No tumor type will be given priority over another and there is no minimum number of glioma patients or solid tumor patients that must be enrolled on the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): The dose level corresponds to 80% of the maximum tolerated dose of LAM561 in adult patients when adjusted for body surface area. The escalation will be to the 100%, and 120% of the maximum tolerated dose of LAM561 in adult patients when adjusted for body surface area. Dose escalation decisions will be made by all active Investigators in collaboration with the Medical Monitor when at least three patients have completed the DLT observation period (Cycle 1) at each dose level. When the third patient at any given dose level has received 14 days of therapy, an "escalation teleconference" will be scheduled after that patient has completed the DLT observation period (Cycle 1). The decision to progress to the next dose level will be made on the basis of review of all significant LAM561-related toxicities.
  Interventions: Drug: LAM561

INTERVENTIONS:
Drug: LAM561 — Once a patient is allocated a dose of LAM561, they will receive the same dose on a daily basis in treatment cycles of 21 days (3 weeks), which may be repeated without therapy interruption until a criterion for discontinuation (clinical or radiological progression of disease, clinically unacceptable toxicity, or another "general" criterion) is met.
  The starting dose will be 2.8 g/m2 twice daily. If tolerated, doses will be escalated to 3.5 g/m2 twice daily and then to a third dose level of 4.2 g/m2 twice daily. These dose levels correspond to 80%, 100%, and 120% of the maximum tolerated dose of LAM561 in adult patients when adjusted for body surface area. A total of 3 dose cohorts are anticipated for the dose escalation phase of the study, with up to 6 patients enrolled at each dose level according to a standard "3+3" design. During each dose cohort, at least 1 week must elapse between the first and subsequent patients receiving treatment with LAM561.

SUMMARY:
An open label, non-randomized study in pediatric patients with advanced high-grade gliomas and other solid tumors.

The study will be performed in two phases: a dose escalation phase in up to 18 patients following a standard "3+3" design to establish dose-limiting toxicity (DLT) and a "safe" dose of LAM561 followed by an expanded safety cohort of up to 10 patients treated at the Maximum Tolerated Dose (MTD). If the MTD is well tolerated in the expanded safety cohort, that dose becomes the Recommended Phase 2 Dose (RP2D).

Glioma patients and other solid tumor patients (including non-glial brain tumors) will be treated as a single cohort. Patients with either tumor type will be allowed to enroll on the study as positions are made available. No tumor type will be given priority over another and there is no minimum number of glioma patients or solid tumor patients that must be enrolled on the trial.

DETAILED DESCRIPTION:
The dose of LAM561 each patient will receive will depend on the dose cohort into which they are enrolled.

Once a patient is allocated a dose of LAM561 (either in the dose escalation phase or the expanded safety cohort), it is planned that they will continue to receive the same dose on a daily basis in treatment cycles of 21 days (3 weeks), which may be repeated continuously without therapy interruption, until any criterion for discontinuation is met (clinical or radiological progression of disease, clinically unacceptable toxicity, or another "general" discontinuation criterion is met as defined in Section 5.5). In the event of significant gastrointestinal toxicity, the treatment schedule may be modified from continuous dosing to an intermittent regime (e.g. 1 week of dosing followed by 1 week not dosing), except during Cycle 1 of the dose escalation phase.

In the case of toxicity, the dose of LAM561 may be reduced or delayed by no more than 14 days at the discretion of the Investigator. Treatment "holidays" of no more than 14 days are also permitted for reasons other than toxicity, except during Cycle 1 of the dose escalation phase.

Intra-patient dose escalation may be permitted in certain specific circumstances (and only if ≤ Grade 2 toxicity was observed during previous treatment cycles), but toxicity will not be considered for definition of DLT.

It is expected that most patients will receive between one and 6 cycles of LAM561 for a treatment period of 3 to 18 weeks. The treatment period may be extended provided that no DLT has been observed and if in the opinion of the Investigator the patient is showing benefit from treatment with LAM561.

Patients demonstrating clinical benefit from LAM561 will have the option of continuing treatment under compassionate use once the study has concluded.

The first cohort of patients has been concluded, and a DSMB meeting was held on 03 April 2023 to assess the safety information in order to initiate the second cohort. The DSMB concluded the safety findings were supportive of initiation of the second cohort, and the second cohort was initiated.

This second cohort has been concluded and another meeting of the DSMB was held on 17 January 2025 to review the safety information and concluded to commence the third cohort of patients with a new dose of idroxioleic acid (2-OHOA).

ELIGIBILITY:
Inclusion Criteria:

1. Age <18 years
2. Diagnosis: Patients must have a histologically- or cytologically-confirmed advanced solid malignancy that is progressive, recurrent or refractory to standard-of-care treatment, or for which there is no standard therapy. Examples of tumors that lack a standard therapy include, but are not limited to, high-grade glioma, diffuse midline glioma, and diffuse intrinsic pontine glioma. For patients with a radiographic diagnosis of diffuse midline glioma or diffuse intrinsic pontine glioma, histologic or cytologic confirmation of their diagnosis is not required.
3. Timing of therapy:

   * Patients must be enrolled before treatment begins. Treatment must start within 14 days of study enrollment.
   * All clinical and laboratory studies to determine eligibility must be performed within 7 days prior to enrollment unless otherwise indicated in the eligibility section.
4. Patients must have a Lansky or Karnofsky performance status score of ≥ 50%, corresponding to ECOG categories of 0, 1 or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients ≤ 16 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair will be considered ambulatory for the purpose of assessing the performance score.
5. Able to swallow and ingest oral medication or have a NG or G-tube for drug administration
6. Able to undergo adequate tumor imaging, via computerized tomography (CT) or magnetic resonance imaging (MRI) scans or any other standardized tumor assessment method based on tumor type (PET, MIBG, etc) to evaluate disease evolution
7. Adequate hematologic, renal, liver function as demonstrated by laboratory values:

   * ANC ≥ 1,000/ul
   * Hemoglobin ≥8.0 gm/dl
   * Platelet count ≥ 100,000/ul
   * Adequate Liver Function Defined As

     * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age, and
     * SGPT (ALT) < 2.5 x upper limit of normal (ULN) for age.
8. Adequate Renal Function Defined As Either

   * Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73m2
   * or a serum creatinine less than or equal to the institutional normal for age
9. No history of QTc prolongation, and a normal QTc interval at screening/baseline (QTc ≤450 msec)
10. No evidence of a bleeding diathesis
11. Negative pregnancy test in women of childbearing potential within 7 days of initiating investigational therapy
12. Patient or legal guardian must give written, informed consent or assent (when applicable) -
13. Recent mothers must agree not to breast feed while receiving medications on study.

Exclusion Criteria:

1. Age ≥ 18 years
2. Known hypersensitivity to any component of the study drug
3. Use of any other investigational drug within five half-lives of that drug prior to the first dose of LAM561
4. Any National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE version 4.0) >Grade 1 toxicities from prior chemotherapy or radiotherapy that could impact on safety outcome assessment
5. Any surgery within 14 days prior to the first dose of LAM561 (excluding shunt or line insertion)
6. Known >Grade 1 intracranial or intratumoral hemorrhage either by CT or MRI scan within the last 1 month. Patients with resolving hemorrhage changes, punctuate hemorrhage or hemosiderin may enter the study
7. A history of significant or uncontrolled cardiovascular disease, including New York Heart Association Class III-IV heart failure, a left ventricular ejection fraction which is clinically significantly abnormal as measured by 2-dimensional (2-D) echocardiogram or Multi Gated Acquisition(MUGA) scan, unstable angina or myocardial infarction within the preceding 6 months
8. Known impairment of gastrointestinal (GI) function that could alter the absorption of study drug (e.g. active Crohn's disease, malabsorption syndrome or states, unresolved diarrhea, small bowel resection or gastric by-pass surgery)
9. Patients who are unable to take oral medications because of significant uncontrolled vomiting will be excluded.
10. A history of uncontrolled hyperlipidemia and/or the need for concurrent lipid lowering therapy
11. Concurrent severe and/or uncontrolled other medical disease (e.g. uncontrolled diabetes mellitus, active uncontrolled infection) that could compromise participation in the study
12. Need for warfarin, phenytoin or sulphonylureas (glibenclamide, glimepiride, glipizide,glyburide or nateglanide)
13. Any serious and/or unstable pre-existing medical, psychiatric or other condition which in the Investigator's opinion could interfere with subject safety, obtaining written informed consent, or compliance with the study protocol
14. Pregnant female patients are not eligible for this study. Pregnancy tests with a negative result must be obtained in all post-menarchal females.
15. Lactating females must agree they will not breastfeed a child while on this study.
16. Males and females of reproductive potential may not participate unless they agree to use an effective contraceptive method and continue to do so for at least 6 months after the completion of therapy.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of LAM561 | Between 1 to 6 cycles (each cycle is 3 weeks)
  To determine the safety and tolerability of LAM561 in pediatric patients (under 18 years) when administered orally using a continuous dosing schedule.
  It will be evaluated through the adverse events [AEs], physical examinations and vital signs, laboratory safety tests and 12-lead electrocardiograms [ECGs].
To identify the Recommended Phase 2 Dose (RP2D) of LAM561 in pediatric patients | Between 1 to 6 cycles (each cycle is 3 weeks)
  The RP2D of LAM561 in pediatric patients will be the Maximum Tolerated Dose during the safety cohort and it's well tolerared.

SECONDARY OUTCOMES:
Characterize LAM561 PK profile | During cycles 1 (Days 1, 8 and 15) and 2 (Day 1) (each cycle is 3 weeks) and at the end of study visit (30 days of the last LAM561 dose)
  The maximum plasma drug concentration observed
Characterize LAM561 PK profile | During cycles 1 (Days 1, 8 and 15) and 2 (Day 1) (each cycle is 3 weeks) and at the end of study visit (30 days of the last LAM561 dose)
  The time at which the maximum plasma concentration is observed
Characterize LAM561 PK profile | During cycles 1 (Days 1, 8 and 15) and 2 (Day 1) (each cycle is 3 weeks) and at the end of study visit (30 days of the last LAM561 dose)
  The area under the plasma concentration versus time curve from time zero to the last quantifiable sampling point, AUC0-t, calculated by using the linear trapezoidal method
Characterize LAM561 PK profile | During cycles 1 (Days 1, 8 and 15) and 2 (Day 1) (each cycle is 3 weeks) and at the end of study visit (30 days of the last LAM561 dose)
  Accumulation ratio (R Cmax). Accumulation ratio calculated from Cmax after repeat dosing and Cmax after single dosing
Characterize LAM561 PK profile | During cycles 1 (Days 1, 8 and 15) and 2 (Day 1) (each cycle is 3 weeks) and at the end of study visit (30 days of the last LAM561 dose)
  Accumulation ratio (R AUC0-t) Accumulation ratio calculated from AUC(0-t) after repeat dosing and AUC(0-t) after single dosing
To assess the preliminary anti-tumor efficacy of LAM561 | Screening and every four cycles (12 weeks)
  Efficacy will be assessed by radiological response of the tumor to treatment

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Arkansas Children's Research Institute, Little Rock, Arkansas
  - University of Miami Hospital, Miami, Florida
  - Hackensack Meridian Health, Inc, Edison, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided